CLINICAL TRIAL: NCT07001020
Title: Innovating Technology Solutions for Residents in Supportive Housing Communities With SUD Through Community-Engaged Research
Brief Title: Innovating Technology Solutions for Residents in Support Housing Communities w SUD Through Community-Engaged Research
Acronym: HousingSUD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Research Behavioral Intervention Strategies, Inc. (Industry)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: DA060718-01; 1R43DA060718-01 (NIH)
Record Dates: First submitted 2025-05-21; First posted 2025-06-03 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Housing Problems; Household Substance Abuse; Substance Use Disorders; Harm Reduction
Keywords: eviction, housing stability, training
MeSH Terms: conditions — Substance-Related Disorders; Harm Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): All participants will be assigned to the intervention, which includes exposure to the technology-based solution while participants are housed within permanent supportive housing. It is anticipated that the intervention will deliver a total of 10 sessions of harm reduction focused cognitive behavioral skills and skills applications. A total of 20 skills practice sessions are also included. Financial incentives are provided up to $50 for completion of sessions and skills practice.
  Interventions: Behavioral: Technology-based Intervention

INTERVENTIONS:
Behavioral: Technology-based Intervention — Technology-based intervention co-developed by a community board.

SUMMARY:
The goal of this clinical trial is to understand whether a technology-based solution, provided to residents in permanent supportive housing, is acceptable, feasible to implement, and has promise for improving resident stability. The main questions it aims to answer are:

• Is the technology-based, community-defined solution usable, acceptable, feasible, and have promise of effectiveness for improving resident knowledge?

There is no comparison group, all participants will receive the technology-based intervention. Researchers expect the intervention will include 2 weeks of intervention content that includes videos and incentives for completing content though the solution tested will ultimately be co-defined by our community board.

DETAILED DESCRIPTION:
Our clinical trial is a pre-post assessment of resident knowledge.

ELIGIBILITY:
Residents:

1. 18 and older;
2. past or current resident in supportive housing community;
3. past or current elevated substance use

Staff:

1. 18 or older;
2. staff at partner agency

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Knowledge | baseline; 30 days
  Knowledge is gain in knowledge related to Cognitive Behavioral Therapy (CBT) skills and life skills taught by the intervention as the number of items answered correctly.
Self-efficacy | baseline; 30 days
  Self-efficacy will assess participant confidence in their ability to implement the skills learned from the intervention. We will develop the items as part of the study, and items will be identified based on the CBT principles and skill applications taught in the program. We will use a 5-point Likert scale of not at all confident (=1) to very confident (=5). A mean score will be computed, ranging from 1 to 5, with higher scores indicating greater self-efficacy in implementing the skills learned in the intervention.
Behavioral intentions | baseline; 30 days
  Behavioral intentions are participants' self-reported likelihood of implementing the skills learned from the intervention on a regular basis. We will develop the items as part of the study, and items will be identified based on the CBT principles and skill applications taught in the program. We will use a 5-point Likert scale of not at all likely (=1) to very likely (=5). A mean score will be computed, ranging from 1 to 5, with higher scores indicating a greater likelihood of implementing the skills learned in the intervention on a regular basis.

OTHER OUTCOMES:
Dosage | Through study completion, an average of 1 month
  Dosage is the number of sessions and skills practices a participant completes

CONTACTS AND LOCATIONS:
Overall Officials: David R Smith, PhD, Principal Investigator — Oregon Research Behavioral Intervention Strategies, Inc.
Locations (1):
- Oregon Research Behavioral Intervention Strategies, Inc., Springfield, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be collected from 25 participants, generating 1 dataset with two assessment time points (baseline, 1-month post-enrollment) including information on participant demographics, knowledge, self-efficacy, and planned behavior. Raw data will be transformed using SPSS and used for statistical analysis. Participant identities, and individual de-identified data will be made available for sharing.
  All quantitative experimental data produced during the course of the project will be preserved and shared.
  To facilitate interpretation of the data, a data dictionary, statistical analysis plans, and data collection instruments will be created, shared, and associated with the relevant datasets.
  Aggregate clinical trials data from all arms of the study will be available in clinicaltrials.gov, along with related metadata. All other data described above in the "data to be shared" section will be deposited into the openICPSR repository.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Shared data generated from this project will be made available as soon as possible, and no later than the time of publication or the end of the funding period, whichever comes first. The duration of preservation and sharing of the data will be a minimum of 5 years after the end of the funding period.
Access Criteria: Survey data will be made available in csv format and will not require the use of specialized tools to be accessed or manipulated.